CLINICAL TRIAL: NCT00347230
Title: Intacs for Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R419/14/2005
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2005-09

CONDITIONS: Keratoconus
Keywords: Intacs ring segments; Keratoconus
MeSH Terms: conditions — Keratoconus

INTERVENTIONS:
Device: Intacs intracorneal ring insertion for the treatment of keratoconus

SUMMARY:
To study the effects Intacs intracorneal ring segments(Addition Technology, Inc) insertion in the treatment of keratoconus

DETAILED DESCRIPTION:
The purpose of this evaluation is to study the effects of implanting INTACS inserts, identical to those commercially available to correct myopia, into the corneal stroma of patients with keratoconus (mild to moderate) and having a clear cornea. The principle of the procedure is to flatten the cornea deformed by keratoconus. One or two segments of the same or a different thickness will be selected to reduce the asymmetric astigmatism responsible for the patient impaired visual acuity.

The surgical technique is based on locating the INTACS inserts on the flattest axis of the refractive error, making the incision on the steepest axis, using 150 degree arc length inserts with different sizes (0.250, 0.300, 0.350, 0.400 & 0.450 mm) according to a nomogram designed for this technique using the INTACS Instrumentation (10-Step Prolate System instruments).

The corneal lamellar channel creation may be performed using the INTACS instrumentation or using the Femtosecond laser (Femtec 20/10 laser[Femtec,Heidelberg Germany])

Primary Assessment Criteria

* Evaluation of the safety of the device for the treatment of patients with keratoconus (mild to moderate)
* Maintenance of best corrected visual acuity (BCVA)
* Improvement in uncorrected visual acuity (UCVA)
* Reduction in manifest refraction spherical equivalent
* Reduction in asymmetric astigmatism

Secondary Assessment Criteria

* Evaluation of the effect of INTACS inserts placement for treatment of corneal ectasia
* Determination of patient satisfaction following the INTACS inserts procedure Patients meeting the eligibility criteria are required to sign a Patient Informed Consent Form prior to study participation.

A thorough examination is perform to evaluate the following:

* Manifest refraction results - Uncorrected visual acuity (UCVA) and best corrected visual acuity (BCVA)
* Cycloplegic refraction results - Uncorrected visual acuity (UCVA) and best corrected visual acuity (BCVA)
* Corneal topography
* Pachymetry
* Step axis location
* Location of incision placement
* Subjective feedback about quality of vision (Excellent, Good, Fair and Poor)

Post-operative Assessment(at 1 day, 1 week, 1 month and 3 months postop)

* Uncorrected visual acuity (UCVA) and best corrected visual acuity with manifest refraction(BCVA) at designated time interval
* Cycloplegic refraction results - Uncorrected visual acuity (UCVA) and best corrected visual acuity (BCVA) at designated time interval
* Corneal topography at designated time interval
* Pachymetry at designated time interval
* Subjective visual outcome ratings over time (Excellent, Good, Fair and Poor)
* Report adverse events

ELIGIBILITY:
Inclusion Criteria:

* Patients must have keratoconus (mild to moderate).
* Visual acuity with contact lenses must be better than or equal to (20/40).
* Patients must be intolerant of contact lenses, i.e., they must be unable to wear contact lenses for a whole day.
* Patients will have a corneal thickness of 425 microns at the site of ICRS (INTACS inserts) placement (the thinnest region of the cornea).
* In terms of general health, patients must not have any illnesses posing an immediate threat to life.
* Patients must have provided written informed consent at least one week prior to surgery.
* Patients must over 21 years of age.
* Patients' contact lenses must have been removed at least one week prior to surgery for soft lenses and two weeks prior to surgery for hard lenses.

Exclusion Criteria:

* Positive pregnancy test.
* Breast-feeding.
* History of previous ophthalmologic surgery on the operative eye.
* Patients with corneal stromal disorders.
* Patients with history of herpetic keratitis.
* Patients with retinal disorders.
* Corneal grafts.
* Patients refusing to remove contact lenses one week before surgery for soft lenses and two weeks before surgery for hard lenses.
* Patients with amblyopia (VA <1110 for the contralateral eye).
* Patients with corneal thickness <425 microns.
* Patients with TOP <10 mmHg or >21 mmHg.
* Patients taking part in other biomedical research in the 30 days prior to the start of this study.
* Patients with an uncooperative disposition.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-10

PRIMARY OUTCOMES:
Visual acuity
Refraction
Corneal topography

SECONDARY OUTCOMES:
Patient satisfaction following procedure

CONTACTS AND LOCATIONS:
Overall Officials: Donald TH Tan, FRCS, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Background] Colin J, Cochener B, Savary G, Malet F, Holmes-Higgin D. INTACS inserts for treating keratoconus: one-year results. Ophthalmology. 2001 Aug;108(8):1409-14. doi: 10.1016/s0161-6420(01)00646-7. PMID 11470691
- [Background] Colin J, Cochener B, Savary G, Malet F. Correcting keratoconus with intracorneal rings. J Cataract Refract Surg. 2000 Aug;26(8):1117-22. doi: 10.1016/s0886-3350(00)00451-x. PMID 11008037
- [Background] Siganos D, Ferrara P, Chatzinikolas K, Bessis N, Papastergiou G. Ferrara intrastromal corneal rings for the correction of keratoconus. J Cataract Refract Surg. 2002 Nov;28(11):1947-51. doi: 10.1016/s0886-3350(02)01495-5. PMID 12457667
- [Background] Schanzlin DJ, Asbell PA, Burris TE, Durrie DS. The intrastromal corneal ring segments. Phase II results for the correction of myopia. Ophthalmology. 1997 Jul;104(7):1067-78. doi: 10.1016/s0161-6420(97)30183-3. PMID 9224455
- [Background] Siganos CS, Kymionis GD, Kartakis N, Theodorakis MA, Astyrakakis N, Pallikaris IG. Management of keratoconus with Intacs. Am J Ophthalmol. 2003 Jan;135(1):64-70. doi: 10.1016/s0002-9394(02)01824-x. PMID 12504699